CLINICAL TRIAL: NCT03700190
Title: Developmental Function and Participation in Life and School Activities in Patients With Autism Spectrum Disorder: A Follow-up Study
Brief Title: The Predictors for Activity and Participation in Children With ASD: A Follow-up Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201601949B0
Record Dates: First submitted 2018-05-11; First posted 2018-10-09 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; activity and participation; sensory perception; facial expression; developmental functions; predictors; follow-up study
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Motor Activity; Facial Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Healthy child
- Experimental: Patients with Autism Spectrum Disorder

SUMMARY:
Developmental function and Participation in life and school activities in patients with autism spectrum disorder: A follow-up study

DETAILED DESCRIPTION:
Most ASD studies have explored the body functions and core symptoms in children with ASD by follow-up, but less studies explore the activities and participation by follow-up, especially the changes in different ages. Although studies explore many predictors to predict the activities and participation in children with ASD, but less studies explore sensory perception to predict the activities and participation in children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Autism Spectrum Disorder
* Age 2-18 y/o
* Agree to sign informed consent

Exclusion Criteria:

* Active medical condition (e.g. infection)
* Concurrent progressive or degenerative disease (e.g. neurogenerative disease)
* Concurrent illness or disease not typically associated with ASD (e.g. pneumonia)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study is a prospective and follow-up study. Children with Autism Spectrum Disorder and Typical Developmental, aged 2-18 years.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of general developmental for Healthy child and patients with Autism Spectrum Disorder in 6 months and 12 months | baseline, 6 months, 12 months
  Comprehensive Developmental Inventory for Infants and Toddlers
Change from baseline of body function & structures in 6 months and 12 months | baseline, 6 months, 12 months
  Bruininks- Oseretsky Test of Motor Proficiency II short form
Change from baseline of Sensory and Perceptual function in 6 months and 12 months | baseline, 6 months, 12 months
  Sensory Profile:It is composed of 125 projects and is completed by the main caregivers of children. There are 14 sub-projects, which can be divided into three main areas: sensory processing (6 items), adjustment (5 items), and emotional response ( 3 items), the project score is divided into 0, 25, 50, 75, 100% (none, rarely, occasionally, often, almost always)
Change from baseline of Participation in 6 months and 12 months | baseline, 6 months, 12 months
  Children Assessment of Participation and Enjoyment(CAPE): Applicable to children or adolescents between the ages of six and twenty one, through questionnaires through self-reports or interviews, a total of 49 questions, asking children about the activities involved in the past four months (1 point for yes, 0 for no).
Change from baseline of Participation in 6 months and 12 months | baseline, 6 months, 12 months
  Preferences for Activity of Children(APCP): For children between the ages of two and five, the questionnaire model is used to allow parents to circle the level. There are 45 questions in total, so that the case or parent can review the activities in the past 4 months and ask if the child have done this activity (1 point means yes, 0 points means no).
Change from baseline of Visual Perception in 6 months and 12 months | baseline, 6 months, 12 months
  Test of Visual Perceptual Skills-Third Edition

SECONDARY OUTCOMES:
Change from baseline of lower extremity function & structures in 6 months and 12 months | baseline, 6 months, 12 months
  Pediatric Balance Scale:The Pediatric Balance Scale (PBS) is a 14-item measure of functional balance for children, ages 2 to 13 years. It was developed through modifications of the Berg Balance Scale to identify children who lack appropriate functional balance and thus may be at risk for developmental delay and injury. The PBS is also used to identify change in functional balance with intervention. The score for each item is from 0 (lowest function) to 4 (highest function). The total maximum score that refers to the best function, is 56.
Change from baseline of activities in 6 months and 12 months | baseline, 6 months, 12 months
  Functional Independence Measure for Children:Applicable to infants and adolescents. The main purpose is to understand and track children's life function performance, progress and goal achievement. There are three main areas: self-care, mobility, and cognition. The score is from 1 to 7 points, 1 is completely dependent, and 7 is completely independent.
Change from baseline of Quality of Life in 6 months and 12 months | baseline, 6 months, 12 months
  TNO-AZL Child Quality of Life Questionnaire (TACQOL): The TACQOL is for children aged from 8 to 15. The questionnaire can be done by the parents or the children themselves for children's health status. The TACQOL contains 56 items with 7 domains (physical functioning, motor, autonomous, cognitive, social, positive moods, and negative moods). There are 8 items in each domain. For physical functioning, motor, autonomous, cognitive and social domains, the scoring is from 0 (never) to 3 (often), followed by a question of child's feeling (3: fine, 2: not so good, 1: quite bad or 0: bad). Items are scored by assigning a value of 4 to the 'never' response, a value of 3 to a 'feeling fine' response, a value of 2 to a 'feeling not so good' response, a value of 1 to a 'feeling quite bad' response and a value of 0 to a 'feeling bad' response. For moods, the scoring is from 0 (never) to 3 (often). The minimal score is 0, and the maximal score is 219.
Change from baseline of Personal & Environment factor in 6 months and 12 months | baseline, 6 months, 12 months
  Parenting Stress Index:Screening and triage measure for evaluating the parenting system and identifying issues that may lead to problems in the child's or parent's behavior. Focuses on three major domains of stress: child characteristics, parent characteristics and situational/demographic life stress.
Change from baseline of Rehabilitation & community service factor in 6 months and 12 months | baseline, 6 months, 12 months
  Measure of Processes of Care: It is to assess parents' perceptions of the care they and their children receive from children's rehabilitation treatment centers. It is a means to assess family-centered behaviors of health care providers. There are 20 items. For each item, a question begins with "To what extent do the people who work with your child," with a 7-point scale with the statement "the service provider engaged in this behavior to a very great extent" (7 point) and "not at all" (1 point). 0 point refers to "not applicable. For each item, the minimal score is 0, and the maximum is 7. A scale score is obtained by calculating the average of the items' ratings. There is no total score.
Change from baseline of Social Responsiveness Scale in 6 months and 12 months | baseline, 6 months, 12 months
  his scale is suitable for children aged 4-18. It is evaluated by 65 questions whether there is a social disorder. The child is identified as autism. The score is 0-3, 0 is untrue, and 3 is descriptive.
Change from baseline of facial expression in 6 months and 12 months | baseline, 6 months, 12 months
  Taiwanese facial expression database:According to Yangming University database, select black and white pictures, strong expression versions, and select five questions of happiness, anger, sadness, fear, and neutrality, a total of 20 questions, each question is taken in four ways, each emotion is in each question will only appear at most, and will be randomly distributed and presented on the computer. The child will specify the specified mood, 1 point for each question, up to 20 points.
Change from baseline of Clancy Behavior Scale in 6 months and 12 months | baseline, 6 months, 12 months
  This scale is suitable for children aged 2-5, a total of 14 questionnaires, about 10 minutes of test, mainly used to screen children with autism, three-point scoring, 2 points for frequent, 1 for occasional, 0 for No, the total score is greater than 14 and there is a tendency to autism. If the score is more than 2/3, it is established as a child with autism.
Change from baseline of Theory of Mind Inventory-2 in 6 months and 12 months | baseline, 6 months, 12 months
  A questionnaire for assessing children's social cognition ability, which is a five-point questionnaire for continuity. It can be filled out by parents or filled by children with good reading skills and speaking skills. This scale is suitable for children aged 2-13, including 60 items. Each question is described as a state, including emotional cognition, mental state understanding, pragmatics and other fields. The person who fills the document is marked with "not", "may not "undetermined", "may have", "determined"
Change from baseline of Childhood Autism Rating Scale II in 6 months and 12 months | baseline, 6 months, 12 months
  Applicable to children under the age of six and those with insufficient intelligence or suspected communication at the age of six, used to judge whether children have autism. A total of 15 questions, each topic is divided into 1 to 4 points, the highest total score of 60 points. For high-function groups, the total score <27.5, non-autistic; between 28 and 33.5 points, there is a tendency to autism; >33.5 points, there is autism.
Change from baseline of Childhood Asperger Syndrome Test in 6 months and 12 months | baseline, 6 months, 12 months
  This is a set of questionnaires for screening autism traits (social impairment, communication deficit, repetitive behavior) for children with Asperger or high-functioning autism. It is suitable for children aged 4-11 years. The questionnaire is filled out by parents and filled out. The time is about 10 minutes, divided into two points (0, 1 points), a total of 37 questions

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, MD, PhD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No